CLINICAL TRIAL: NCT03826706
Title: Comparison Of Storz C-Mac® D Blade Videolaryngoscope With McGrath® X3 Blade Videolaryngoscope In Double Lumen Tube Patients
Brief Title: Comparison Of Videolaryngoscopes In Double Lumen Tube
Acronym: D&Xblade
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Ahmet Selim Ozkan, Asst. Prof. Dr. Ahmet Selim Ozkan, Inonu University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: Asozkan 4
Record Dates: First submitted 2019-01-30; First posted 2019-02-01 (Actual); Last update posted 2019-02-05 (Actual); Status verified 2019-02

CONDITIONS: Videolaryngoscopy; Double Lumen Tube; One-lung Ventilation
Keywords: Videolaryngoscopy; Double lumen tube; One-lung ventilation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- C-MAC Videolaryngoscope D blade (Active Comparator): Patients was intubated with C-MAC videolaryngoscope D blade.
  Interventions: Device: C-MAC Videolaryngoscope D blade; Device: McGrath MAC Videolaryngoscope X3 blade
- McGrath MAC Videolaryngoscope X3 blade (Active Comparator): Patients was intubated with McGrath MAC Videolaryngoscope X3 blade
  Interventions: Device: C-MAC Videolaryngoscope D blade; Device: McGrath MAC Videolaryngoscope X3 blade

INTERVENTIONS:
Device: C-MAC Videolaryngoscope D blade — C-MAC videolaryngoscope D blade An intubating device that is used for endotracheal intubation. Endotracheal intubation was applied by anesthesiologist with C-MAC videolaryngoscope.
Device: McGrath MAC Videolaryngoscope X3 blade — McGrath MAC videolaryngoscope X blade An intubating device that is used for endotracheal intubation. Endotracheal intubation was applied by anesthesiologist with McGrath MAC videolaryngoscope.

SUMMARY:
Along with the technological advances in medicine, videolaryngoscope is the most commonly preferred technique for intubation with double lumen tube. The use of Storz C-MAC D Blade and McGrath MAC X3 Blade videolaryngoscope were compared in intubation of single lung ventilation patients who underwent chest surgery in terms of duration of intubation, hemodynamic response and intubation-induced complications.

DETAILED DESCRIPTION:
It is very important for anesthesiologists to evaluate and make the airway safe in order to start and continue surgical operations. Endotracheal intubation has many important reasons such as ensuring airway control safely during surgical procedure, increasing the depth of anesthesia, need interventions for surgical or anesthetic complications, reduction of dead space, reduction of respiratory effort and prevention of aspiration risk. Videolaryngoscope, developed in recent years and beginning to take place in the algorithms, facilitate difficult airway management and hence intubation.

The use of videolaryngoscope in patients with intubation such as double lumen tube, has been frequently reported in the literature. McGrath videolaryngoscope has a high-resolution video camera, a length-adjustable angle blade, and a light source at the tip of the blade. At the same time, the C-MAC videolaryngoscope is another advanced videolaryngoscope with a better quality video and camera system and improves the performance of videolaryngoscope with some technological changes. In this prospective controlled clinical study, the purpose is to compare C-MAC videolaryngoscope with D blade and McGrath MAC videolaryngoscope with X3 blade in respect to duration of intubation, haemodynamic response, and adverse events associated with intubation of patients undergoing lung surgery.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiology score III,
* 18-65 years,
* BMI> 40
* Patients who was intubated with double lumen tube.

Exclusion Criteria:

* American Society of Anesthesiology IV,
* Under 18 years,
* Over 65 years,
* Under BMI<40
* Obstetric patients,
* Uncontrolled cerebrovascular disease,
* Patients who refused written informed consent forms

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-02-15 (Estimated); Primary Completion 2019-03-30 (Estimated); Study Completion 2019-04-10 (Estimated)

PRIMARY OUTCOMES:
Time to intubation | From beginning of holding videolaryngoscope to seeing two meaningful end-tidal carbon dioxide levels up to 3 minutes
  Time to intubation was defined as the time from when the anesthesiologist picked up the videolaryngoscope to when the anesthesiologist successfully placed the endotracheal tube through the vocal cords

SECONDARY OUTCOMES:
Heart Rate | From beginning of Anesthesia induction to 5th minutes of intubation
  Heart Rate
Mean Arterial Pressure | At beginning of Anesthesia induction, 1st, 2nd, 3th and 5th minutes of intubation
  Mean Arterial Pressure
Adverse Events | During the first 24 hour postoperatively
  Bleeding in the mouth, edema in the mouth, burst of intubation tube cuff, external laryngeal press, presence of head position change, laryngospasm, hypoxia, hoarseness, throat ache

CONTACTS AND LOCATIONS:
Overall Officials: Ahmet Selim Ozkan, Study Director — Inonu University Medical Faculty
Locations (1):
- Ahmet Selim Ozkan, Malatya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No